CLINICAL TRIAL: NCT02790983
Title: Primary Tumor Research and Outcomes Network (PTRON) A Multicenter Prospective Registry for the Management and Outcomes of Primary Tumors of the Spine
Brief Title: Primary Tumor Research and Outcomes Network
Acronym: PTRON
Status: Recruiting | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Collaborators: AO Foundation, AO Spine (Other)
Responsible Party: Sponsor
Other Study IDs: PTRON
Record Dates: First submitted 2016-05-18; First posted 2016-06-06 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Spinal Column Tumor
Keywords: Registry; Spine; Surgery; Medical Oncology; Radiation Oncology; Neoplasms; Systemic Oncologic Therapy; Radiation Therapy; Tumor Markers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Tumor tissue and adjacent normal tissue Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
This project aims to establish a network of spine oncology centers dedicated to prospective multicenter research of patients diagnosed with a primary tumor of the spine and will include a comprehensive prospective clinical database which will serve as a shared research platform. Demographic, clinical, diagnostic, and therapeutic variables will be used to answer questions about survival and local recurrence, as well as questions about adverse events (AEs), morbidity data, and health-related quality of life (HRQOL) outcomes.

DETAILED DESCRIPTION:
Objective: To prospectively investigate variables (clinical, diagnostic, and therapeutic) in patients diagnosed with primary spinal column and cord tumors that are associated with:

* survival
* local recurrence
* morbidity data
* patient reported outcomes

Outcome measures: Variables applicable to primary spinal column tumor patients which will be collected in the registry include:

* Patient details
* Treatment status
* Details of previous treatment
* Diagnosis and biopsy types
* Tumor details
* Oncological staging
* Symptoms
* Treatment details
* Imaging information

We aim to collect the following outcome measures:

* Overall survival data
* Local disease recurrence data
* Morbidity data
* Patient reported outcomes:
* Euroquol-5D-3L, EQ-5D-Y (if applicable)
* Euroquol EQ-5D VAS - Quality of Life
* Neck pain numeric rating scale (NRS)
* Arm pain NRS
* Back pain NRS
* Leg Pain NRS
* SF-36 version 2
* SOSG Outcome Questionnaire (SOSGOQ) v1.0 and v2.0
* Surverys on patient expectations and satisfaction

ELIGIBILITY:
Inclusion criteria

* Patient with a current primary spine tumor or history of a primary spine tumor, including tumors within or surrounding the spinal column and/or spinal cord. This includes extradural tumors, intramedullary tumors (i.e. astrocytomas, ependymoma, etc.) and extramedullary tumors (i.e. meningiomas, neurofibromas, schwannomas, etc.).
* Informed consent obtained, i.e.:

  * Ability to understand the content of the patient information/ICF
  * Willingness and ability to participate in the registry according to the Registry Plan (RP)
  * Signed and dated EC/IRB approved written informed consent

OR

* Written consent provided according to the IRB/EC defined and approved procedures for patients who are not able to provide independent written informed consent

Exclusion Criteria:

- Patient diagnosed with a metastatic tumor of the spine.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with a primary tumor of the spine or patients with a history of a spine tumor
Sampling Method: Non-Probability Sample
Enrollment: 1350 (Estimated)
Dates: Start 2016-10; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival data | From the date of enrollment until the date of dropout (ie. consent withdrawal, lost-to follow-up or death) which can be up to 25 years
  FU visits will be scheduled and performed according to the local standard of care and at each scheduled visit the patient's survival will be documented. In case a patient misses a scheduled visit it will be assessed if the patient is still alive
Local disease recurrence data | From the date of enrollment until the date of dropout (ie. consent withdrawal, lost-to follow-up or death) which can be up to 25 years
  At first prospective treatment and every FU visit, each patient, regardless of which stage they are at in their treatment, will be evaluated for local disease recurrence. Patients that are classified as "non-virgin" will be evaluated for local disease recurrence also at baseline.
Perioperative morbidity data | From the date of enrollment until the date of dropout (ie. consent withdrawal, lost-to follow-up or death) which can be up to 25 years
  Complications will be assessed by evaluating the patient's medical files from the time treatment was initiated until the day of follow-up.
  Intraoperative complications: (Airway/ventilation; Allergic reaction; Anesthesia related; Bone implant interface failure requiring revision; Cardiac; Cord injury; Dural tear; Hardware malposition requiring revision; Hypotension ; Massive blood loss ; Nerve root injury; Pressure sores; Vascular injury; Visceral injury; Other).
  Pre-/post treatment complications: (Cardiac arrest/failure/arrhythmia; Construct failure with loss of correction; Construct failure without loss of correction; CSF leak/meningocele; Deep vein thrombosis; Deep wound infection; Delirium; Dysphagia; Dysphonia; GI bleeding; Hematoma; Myocardial infarction; Neurologic deterioration; Non-union; Pneumonia; Postoperative neuropathic pain; Pressure sores; Pulmonary embolism; Superficial wound infection; Systemic infection; Urinary tract infection; Wound dehiscence; Other)

SECONDARY OUTCOMES:
Euroqol EQ-5D-3L or Euroqol EQ-5D-Y (for patients <16y) | From the date of enrollment until the date of dropout (ie. consent withdrawal, lost-to follow-up or death) which can be up to 25 years
  The EuroQOL group developed a standardized instrument for use as a measure of health outcome. Applicable to a wide range of health conditions and treatments, it contains 5 questions and provides a simple descriptive profile and a single index value for health status.
  EQ-5D is designed for self-completion by respondents and is ideally suited for use in mailed surveys, in clinics and face-to-face interviews. It is cognitively simple, taking only a few minutes to complete. Instructions to respondents are included in the questionnaire.
Pain Numeric Rating Scale | From the date of enrollment until the date of dropout (ie. consent withdrawal, lost-to follow-up or death) which can be up to 25 years
  It will be assessed for neck, back, leg and arm. The Pain NRS is an 11-point horizontal scale where the end points are the extremes of no pain (0) and pain as bad as it could be, or worst pain (10). It measures subjective intensity of pain and the patient rates his/her overall or average daily pain.
SF-36 version 2 | From the date of enrollment until the date of dropout (ie. consent withdrawal, lost-to follow-up or death) which can be up to 25 years
  It is a multipurpose, short-form health survey with 36 questions. It yields an eight-scale profile of scores: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions. In addition, two composite scores are constructed using factorial modeling, one for physical health (Physical Composite Score - PCS) and one for mental health (Mental Composite Score - MCS). A scoring algorithm is available using linear T-score transformation that translates scores using population based norms into scores with mean = 50 and standard deviation = 10. The algorithm is available for all 8 subscales as well for the PCS and MCS.
Spine Oncology Study Group Outcome Questionnaire | From the date of enrollment until the date of dropout (ie. consent withdrawal, lost-to follow-up or death) which can be up to 25 years
  This is a new HRQOL outcome tool which was developed specifically for metastatic spine disease. It is currently available in English and Hungarian. It contains 20 items representing all four domains of the International Classification of Function and Disability. Additionally, there are seven follow-up questions referring to treatment satisfaction. It is made up of five domains: physical function, neural function, pain, mental health, and social function. During the first phase of this registry, patients completed the SOSGOQ version 1.0. The English SOSGOQ version 2.0 was released in January 2018 and will be used
Survey on patient expectation | Prior to surgical treatment
  A survey on the patient's expectation regarding the surgery. Only applicable for patients that receive surgical treatment.
Survey on patient satisfaction | After surgical treatment until the date of dropout (ie. consent withdrawal, lost to follow-up or death) which can be up to 25 years
  A survey on the patient's satisfaction post-surgery. Only applicable for patients that receive surgical treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Reynolds, MD, Principal Investigator — Clinical Lead for Spinal Surgery at Oxford University Hospitals
Locations (19):
- United States (9):
  - University of California, Los Angeles, California
  - UCSF Medical Center, San Francisco, California
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Rhode Island Hospital, Providence, Rhode Island
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
- University of Queensland, School of Medicine, Brisbane, Australia
- Canada (2):
  - Vancouver General Hospital and the University of British Columbia, Vancouver, British Columbia
  - Toronto Western Hospital, Toronto, Ontario
- Peking University 3rd Hospital, Beijing, Beijing Municipality, China
- Universitaetsklinikum Carl Gustav Carus der Techn. Universitaet - Dresden, Dresden, Germany
- National Center for Spinal Disorders and Buda Health Center, Budapest, Hungary
- Italy (2):
  - Istituto Ortopedico Rizzoli, Bologna
  - IRCCS Istituto Ortopedico Galeazzi, Milan
- Kanazawa Medical University Hospital, Kanazawa, Japan
- Oxford University Hospitals, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No